CLINICAL TRIAL: NCT05957874
Title: The Effect of Sleep Hygiene Training Implemented With the Combined Package Program on Sleep Deprivation and Sleep Habits in Children
Brief Title: The Effect of Sleep Hygiene Training Implemented
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Semra Kose, Asisstant Proffessor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NEUSKose1
Record Dates: First submitted 2023-07-09; First posted 2023-07-24 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Sleep Hygiene
Keywords: Sleep; sleep deprivation; sleep habit; nurse; school-age children
MeSH Terms: conditions — Sleep Hygiene; Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: This study is an experimental study with pretest and posttest control measurement and control group.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental): Questionnaires will be applied to the children and their families who agree to participate. A one-week sleep hygiene training will be given for three consecutive days. On the first day of education, children will be given a checklist and tasks that will facilitate the transition to weekly sleep. In addition, within the scope of using technology positively, reminders including sleep hygiene principles will be sent to families every day for four weeks via a social media tool. Total intervention time is planned as 4 weeks. The researchers planned to start the trainings on Monday. At the beginning of each week, face-to-face interviews will be held with the students in the experimental group and it will be evaluated whether the tasks have been fulfilled. At the end of 4 weeks, the final test application of the experimental group will be made. Then, the questionnaires will be applied again after 2 weeks for control measurement.
  Interventions: Other: Combined package program
- Control (No Intervention): The children who agreed to participate in the class determined as the control group as a result of drawing lots and the children and their families who agreed to participate will fill in the "Sociodemographic Characteristics and Introductory Information Form", the "Sleep Deprivation Scale for Children and Adolescents" and the mothers will fill in the "Child Sleep Habits Questionnaire". At the end of 4 weeks, the post-test application of the control group will be made. After the tests are applied, training will be given to the control group on a suitable day for the class and the training booklet will be distributed.

INTERVENTIONS:
Other: Combined package program — Combined package program content:
  * Training: A one-week sleep hygiene training will be given to the experimental group. The training will take an average of 30 minutes for three consecutive days and a training booklet will be provided. In addition, two posters will be prepared to hang in the classroom. In one of the posters, a sleep hygiene rule will be placed at each hour using the clock order. In the other poster, good and bad sleep habits will be placed in the form of do-do.
  * Task Flower: Tasks that will facilitate the transition to weekly sleep will be given to the children of the experimental group. Tasks are applications to be done within 30-60 minutes before going to bed. After the tasks, the children will perform their daily sleep routine and go to sleep.
  * Notifications: As part of using technology positively, reminders will be sent to families every day for two weeks via a social media tool. These warnings will include sleep hygiene principles.
  Arms: Experiment

SUMMARY:
Good and quality sleep, which has an important place in the lives of all living things; important for the health and well-being of children. Proper sleep habits are needed for quality and adequate sleep. According to the National Sleep Foundation, these habits include practices such as regular bedtimes, sleep routines, screen restrictions before bed. With the age of starting school in children; Due to the roles brought by school, lessons and social obligations, problems such as delay in bedtime and shorter sleep time are seen. Shortening of sleep time causes sleep deprivation. sleep deprivation; It is defined as a delay in bedtime and a shorter sleep time than would normally be due to intentional or daily activities. The use of sleep hygiene interventions to address sleep deprivation in children is highly effective. Sleep hygiene is a cost-effective method that is performed without the need for any additional material, consisting of both environmental and behavioral habits. In our study, a quasi-experimental pretest-posttest-control study design with a control group will be used to determine the effect of sleep hygiene education applied with the combined package program on sleep deprivation and sleep habits in children. After the necessary permissions are obtained, the classes will be divided into experiments and controls by drawing lots. To the experimental group; After the pre-test is applied, training and tasks will be given. In addition, a sleep hygiene policy will be sent to the families by phone every day. The total intervention will last four weeks, at the end of which a post-test will be administered. Two weeks will be waited without intervention, two weeks later the control measurement will be made. To the control group; Pre-test and post-test will be applied at the same time with the experimental group and training will be given after the post-test. The research data will be evaluated with the Statistical Package for the Social Sciences (SPSS) statistical program on the computer and in the form of numbers, percentages, averages and standard deviations for descriptive statistics in the computer environment and with necessary statistical analyzes. Significance will be accepted as p<0.05 at α=95% confidence interval.

DETAILED DESCRIPTION:
Sleep; It is a physiological need that has a very strong effect on increasing the quality of life of individuals. Good and quality sleep for children, which has an important place in the lives of all living things; important for their health and well-being. in children; ensuring healthy growth and development, establishment of homeostatic balance mechanism, sensory and hormonal development, improvement of metabolism and immune system, cognitive development, memory, academic performance, cardiovascular risk, obesity; Psychological conditions such as depression, suicidality, paranoia, and hallucinations have been associated with sleep quality and adequacy.

Proper sleep habits are needed for quality and adequate sleep. According to the National Sleep Foundation, these habits include practices such as regular bedtimes, sleep routines, screen restrictions before bedtime. A circadian rhythm develops until the age of 6, and after the age of 6, the habit of being a night owl or getting up early is observed. In addition, with the school starting age (after the age of 6), children enter into a busy schedule and their sleeping habits may change. Adequate sleep time for school-age children is 9-11 hours.

With the age of starting school in children; Due to the roles brought by school, lessons and social obligations, problems such as delay in bedtime and shorter sleep time are observed. Shortening of sleep time causes sleep deprivation. sleep deprivation; It is defined as a delay in bedtime and a shorter sleep time than it should be, either intentionally or due to daily actions. sleep deprivation in children; It causes decrease in cognitive performance, poor school performance, weakening of mental abilities, daytime sleepiness, lack of physical activity, obesity and changes in dietary habits (short sleep calorie foods and carbonated drink consumption; adequate sleep fruit and vegetable consumption. For these reasons, it is of great importance to eliminate sleep deprivation in children. The use of sleep hygiene interventions to address sleep deprivation in children is highly effective. Sleep hygiene is a set of behaviors that aim to improve sleep quality by eliminating bad sleep habits. Sleep hygiene is a cost-effective method that is performed without the need for any additional material, consisting of both environmental and behavioral habits. It is known that sleep hygiene interventions, especially performed at school, are very effective and applicable.

When the literature is examined, sleep hygiene interventions are generally focused on children with a health problem (hyperactivity, autism, sleep problems, etc. Although the effects of sleep on school performance are known, interventions to improve the sleep quality of healthy school-age children are very few. School is a very effective environment in developing healthy behavior, and the home environment is important for the behavior to continue. For these reasons, in our study, school-age children who do not have any health problems will be handled using both the school environment and the home environment. The research to be carried out is unique from other studies in that it aims to create behavior in children by using the school and home environment together and by attracting the attention of the materials used by the children. As a result of the examinations (yök thesis, google academic Turkish, etc.), our research is the first in Turkey in terms of being aimed at healthy children, the intervention for both children and families, and a quasi-experimental research design.

ELIGIBILITY:
Inclusion Criteria:

* The child is studying in the 4th grade (9-11 years old)
* Ability to read, write and speak Turkish
* The willingness of the family and the child to participate in the research
* Having internet access

Exclusion Criteria:

* Using any sleeping pills
* Presence of a concomitant chronic disease
* Having received any training on sleep
* Existence of a situation that will prevent the understanding of the given education

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2023-07-09 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Sociodemographic Characteristics and Introductory Information Form | 1st week (pretest)
  This form, which was created by the researchers by scanning the literature, also includes age, gender, educational status of parents, sleeping and waking hours, etc. There are 17 questions

SECONDARY OUTCOMES:
Sleep Deprivation Scale for Children and Adolescents | After the pretest in the 1st week, the posttest in the 4th week and the control measurement in the 6th week will be done.
  In the context of the validity and reliability study of the Child and Adolescent Sleep Deprivation Scale developed by Kandemir et al., this form was created regarding the sleep needs of children and adolescents attending school. The scale can be applied to children and adolescents between the ages of 8-17. The scale, which emerged as a one-dimensional structure, consists of 15 items and a 4-point Likert type prepared as "strongly disagree", "disagree", "agree" and "strongly agree". The Cronbach Alpha value of the scale is 0.94. The lowest score that can be obtained from the scale is 15 and the highest score is 60. As the score from the scale increases, sleep deprivation increases, and as it decreases, sleep deprivation decreases.

OTHER OUTCOMES:
Child Sleep Habits Questionnaire | After the pretest in the 1st week, the posttest in the 4th week and the control measurement in the 6th week will be done.
  The abbreviated form of the Children's Sleep Habits Questionnaire (CSHQ), developed by Owens et al. in 2000, was adapted to Turkish by Perdahlı Fiş et al. The scale is filled by the mothers and/or fathers of primary school 1st, 2nd, 3rd, 4th grade students. The mother and/or father are asked to evaluate the child's sleep habits considering the past week. The scale consists of 33 items. The scale has eight sub-dimensions, which can be listed as bedtime resistance, delayed falling asleep, sleep duration, sleep anxiety, night awakenings, parasomnias, impaired breathing during sleep, and daytime sleepiness. Cronbach's alpha value was found to be 0.78. 41 points obtained from the scale are accepted as the cut-off point, and values above this are considered clinically significant.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan Üniversitesi Hemşirelik Fakültesi, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The decision to share the study results will be made during the study period or when it is concluded.

REFERENCES:
- [Result] Ahmadi, Z., & Omidvar, S. (2022). The quality of sleep and daytime sleepiness and their association with quality of school life and school achievement among students. Journal of Education and Health Promotion, 11(1), 159. https://doi.org/10.4103/JEHP.JEHP_22_22 Åslund, L., Arnberg, F., Kanstrup, M., & Lekander, M. (2018). Cognitive and Behavioral Interventions to Improve Sleep in School-Age Children and Adolescents: A Systematic Review and Meta-Analysis. Journal of Clinical Sleep Medicine: JCSM: Official Publication of the American Academy of Sleep Medicine, 14(11), 1937. https://doi.org/10.5664/JCSM.7498 Bora, I. H. Dr., & Bican, A. Dr. (2007). Sleep Physiology. Journal of Turkish Clinics, 3(23), 1-6. Busch, V., Altenburg, T. M., Harmsen, I. A., & Chinapaw, M. J. (2017). Interventions that stimulate healthy sleep in school-aged children: a systematic literature review. European Journal of Public Health, 27(1), 53-65. https://doi.org/10.1093/EURPUB/CKW140 Córdova, F. V., Barja, S., & Brockmann, P. E. (2018). Consequences of short sleep duration on the dietary intake in children: A systematic review and metanalysis. Sleep Medicine Reviews, 42, 68-84. https://doi.org/10.1016/J.SMRV.2018.05.006 Freeman, D., Sheaves, B., Goodwin, G. M., Yu, L.-M., Nickless, A., Harrison, P. J., Emsley, R., Luik, A. I., Foster, R. G., Wadekar, V., Hinds , C., Gumley, A., Jones, R., Lightman, S., Jones, S., Bentall, R., Kinderman, P., Rowse, G., Brugha, T., … Espie, C. A. (2017 ). Articles The effects of improving sleep on mental health (OASIS): a randomized controlled trial with mediation analysis. The Lancet. Psychiatry, 749. https://doi.org/10.1016/S2215-0366(17)30328-0 Gruber, R., Somerville, G., Bergmame, L., Fontil, L., & Paquin, S. (2016). School-based sleep education program improves sleep and academic performance of school-age children. https://doi.org/10.1016/j.sleep.2016.01.012 Hirshkowitz, M., Whiton, K., Albert, S. M., Alessi, C., Bruni, O., Doncarlos, L., Hazen, N., Herman, J., Katz, E. S., Kheirandish-Gozal, L., Neubauer, D. N., O'donnell, A. E., Ohayon, M., Peever, J., Rawding, R., Sachdeva, R. C., Setters, B., Vitiello, M. V, Catesby Ware, J., & Hillard, P. J. A. (2015). National Sleep Foundation's sleep time duration recommendations: methodology and results summary. Sleep Health, 1, 40-43. https://doi.org/10.1016/j.sleh.2014.12.010 Hiscock, H., Quach, J., Paton, K., Peat, R., Gold, L., Arnup, S., Sia, K. L., Nicolaou, E., & Wake, M. (2018). Impact of a Behavioral Sleep Intervention on New School Entrants' Social Emotional Functioning and Sleep: A Translational Randomized Trial. https://Doi.Org/10.1080/1540202.2018.1469493, 17(6), 698-712. https://doi.org/10.1080/1540202.2018.1469493 İşsever, O., Akçay Didişen, N., & Bal Yilmaz, H. (2021). An Important Topic in Child Care: Safe Sleep and Sleep Education. Journal of Izmir Katip Celebi University Faculty of Health Sciences, 6(2), 157-161. Kandemir, M., Bozdemir, E., Hayran, Y., Tonga, Z., & Kandemir, A. (2021). Sleep Deprivation Scale for Children and Adolescents. Journal of Interdisciplinary Education: Theory and Practice. https://doi.org/10.47157/jietp.875187 Loring, W., & Malow, B. (2022). Sleep Hygiene and Related Interventions: Their Impact on Sleep. Clinical Handbook of Behavioral Sleep Treatment in Children on the Autism Spectrum, 127-136. https://doi.org/10.1007/978-3-030-99134-0_9 Matricciani, L., Paquet, C., Galland, B., Short, M., & Olds, T. (2019). Children's sleep and health: A meta-review. Sleep Medicine Reviews, 46, 136-150. https://doi.org/10.1016/J.SMRV.2019.04.011